CLINICAL TRIAL: NCT05132231
Title: CARE: A CAnadian Real World Evidence Study of Brodalumab in Plaque Psoriasis to Understand the Impact on Quality of Life and Work Productivity
Brief Title: Canadian Real World Evidence Study of Brodalumab in Plaque Psoriasis to Understand the Impact on Quality of Life and Work Productivity
Acronym: CARE
Status: Active, not recruiting | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BHC-CANDerm-003
Record Dates: First submitted 2021-10-22; First posted 2021-11-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Brodalumab initiator: Eligible adult participants who are enrolling into the SILIQ (brodalumab) Patient Support Program (PSP) and initiating brodalumab as per routine care.
  Interventions: Biological: Brodalumab
- Matched cohort: Participants treated with other therapies, with similar characteristics as the subgroup (participants who can be linked to an administrative health services database) of brodalumab treated participants such as age, gender/sex, comorbidities, and prior biologic experience.
  Interventions: Biological: Matched cohort

INTERVENTIONS:
Biological: Brodalumab — Brodalumab
  Groups: Brodalumab initiator
Biological: Matched cohort — Matched cohort
  Groups: Matched cohort

SUMMARY:
This is a phase IV, 12-month observational, prospective, open-label, multi-center study that will be conducted across approximately 50 sites in Canada for an estimated study duration of 32 months. All eligible adult participants who are enrolling into the SILIQ Patient Support Program (PSP) and initiating brodalumab as per routine care may be offered participation in the study. If the participant agrees, their verbal consent and details will be entered into the study platform by the enrolling physician so that the participant can access the electronic informed consent form. Participants who meet the eligibility criteria and provide electronic informed consent will be enrolled in the study. The study observation period will be 12 months (±15 days). Data will be collected on approximately 500 participants across academic and community centers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years old at the time of verbal consent to participate in the study.
2. Initiating brodalumab as part of routine clinical care through the SILIQ (brodalumab) Patient Support Program (PSP) for the treatment of plaque psoriasis but has not yet received their first dose. Decision to treat with brodalumab must have been reached prior to and independently of recruitment in the study.
3. Must be able to read, understand, and communicate in English or French.
4. Willing and able to provide informed consent on an online platform using an Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved electronic Informed Consent Form (ICF) in English or French.

Exclusion Criteria:

1. Not willing or able to complete ePROs (electronic Patient Reported Outcomes) on an online platform (using a computer or mobile device).
2. Participation in brodalumab phase IV study (NCT04149587).
3. Participation in an interventional clinical trial concurrently or within the last 30 days prior to providing verbal consent to participate in this study.
4. Patient with Crohn's disease or with clinically significant hypersensitivity to brodalumab or to any of the excipients or component of the container (contraindications as per the Product Monograph).
5. Presence of any other serious and/or uncontrolled medical condition that, in the opinion of the investigator, prohibits the patient from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants initiating brodalumab as part of routine clinical care and who meet all of the inclusion and none of the exclusion criteria are eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The percentage change from baseline of the Dermatology Life Quality Index (DLQI) at 3 months, 6 months, and 12 months post-brodalumab initiation. | baseline, 3 months, 6 months, 12 months
  The Dermatology Life Quality Index (DLQI) measure is self administered and includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school. Each item has four response categories, ranging from 0 (not at all or not relevant) to 3 (very much) assessing the impact of the disease over the last week. The DLQI total score is a sum of the 10 questions. Scores range from 0 to 30 and higher scores indicate greater health-related quality-of-life impairment.
The percentage change from baseline of the Work Productivity and Activity Impairment: Psoriasis (WPAI:PSO) component scores at 3 months, 6 months, and 12 months post-brodalumab initiation. | baseline, 3 months, 6 months, 12 months
  The Work Productivity and Activity Impairment: Psoriasis (WPAI:PSO) is a validated self-reported 6-item questionnaire that allows quantitative assessment of the effects of PsO on work productivity, daily activities, and classroom impairment. Scores are calculated as percentages of hours worked and percentages of productivity at work on workdays for respondents who are employed at the time of questionnaire completion.
The percentage change from baseline of the Health Utility Index (HUI2) at 3 months, 6 months, and 12 months post-brodalumab initiation. | baseline, 3 months, 6 months, 12 months
  The Health Utility Index (HUI2) is a 15-item questionnaire that allows researchers to classify the health status of patients and consists of seven attributes (sensation, mobility, emotion, cognition, self-care, pain, and fertility). Health state levels for descriptive responses are converted to health utilities scores using single- and multi-attribute utility functions that consist of look-up tables and mathematical formulae. Utility values for HUI2 range from -0.03 to 1.00, where a value of 1.00 indicates perfect health and a score of 0.00 corresponds to death. Negative scores represent health states considered to be worse than death.
The mean Treatment Satisfaction Questionnaire for Medication (TSQM) domain scores at baseline, 3 months, 6 months, and 12 months post-brodalumab initiation. | baseline, 3 months, 6 months, 12 months
  The self-administered Treatment Satisfaction Questionnaire for Medication (TSQM) questionnaire is along 4 dimensions: medication effectiveness, side effects of use, convenience of use, and global/overall satisfaction. The scale for TSQM scores ranges from 0 (extremely dissatisfied) to 100 (extremely satisfied).

SECONDARY OUTCOMES:
The number and percentage of patients on brodalumab at baseline, 3 months, 6 months, and 12 months post-initiation by key patient demographics and clinical characteristics. | baseline, 3 months, 6 months, 12 months
  Key demographics and clinical characteristics include: prior biologic experience, age, gender, province, disease duration, number of comorbidities.
The number and percentage of patients that initiated brodalumab achieving a Psoriasis Area Severity Index (PASI) response of 75, 90 or 100 at 3 months, 6 months, and 12 months post-brodalumab initiation. | baseline, 3 months, 6 months, 12 months
  The Psoriasis Area Severity Index (PASI) score (0 to 72) is a calculation of plaque qualities, including induration/infiltration (plaque thickness), erythema, and desquamation (scaling), and the area involved with PsO (48). The investigator or qualified designee will score plaque erythema, scaling and induration (on a scale of 0 to 4) and area of involvement (on a scale of 0 to 6) for 4 body areas: head and neck, upper extremities, trunk, and lower extremities.
The number and percentage of patients that initiated brodalumab achieving an Static Physicians Global Assessment (sPGA) score of 0 or 1 at 3 months, 6 months, and 12 months post-brodalumab initiation. | baseline, 3 months, 6 months, 12 months
  The Static Physicians Global Assessment (sPGA) scale (0 [clear] to 4 [severe]) is designed to evaluate the assessor's global assessment of the patient's psoriasis.
The number and percentage of patients that initiated brodalumab achieving a 2 grade or more improvement compared to baseline of the Static Physicians Global Assessment (sPGA) score at 3 months, 6 months, and 12 months post-brodalumab initiation. | baseline, 3 months, 6 months, 12 months
  The Static Physicians Global Assessment (sPGA) scale (0 [clear] to 4 [severe]) is designed to evaluate the assessor's global assessment of the patient's psoriasis.
The percentage change from baseline of the Psoriasis Symptom Inventory (PSI) at 3, 6, and 12 months post-brodalumab initiation. | baseline, 3 months, 6 months, 12 months
  Psoriasis Symptom Inventory (PSI): The severity of itch, redness, scaling, burning, stinging, cracking, flaking, and pain over the last 24 hours is assessed on a scale of 0 to 4 (0 - not at all, 1- mild, 2 - moderate, 3- severe, 4- very severe) for a total score of 32, with higher scores indicating more severe disease
The number and percentage of Adverse Events (AEs) or (Serious Adverse Events) SAEs reported over 12 months post-brodalumab initiation. | 12 months
Reasons for discontinuation of brodalumab therapy. | 12 months
  Discontinuation reason is captured on the case report form.
The number and percentage of patients who initiated brodalumab and remained on treatment after 3 months, 6 months and 12 months post-brodalumab initiation. | 12 months
The mean and median time to brodalumab discontinuation. | 12 months
The number of patients encountering psoriasis-related physician | baseline, 3 months, 6 months, 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures.
Associated costs of patients encountering psoriasis-related physician | baseline, 3 months, 6 months, 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures.
The number of patients encountering hospital visit | baseline, 3 months, 6 months, 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures.
Associated costs of patients encountering hospital visit | baseline, 3 months, 6 months, 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures.
The number of patients encountering emergency room (ER) visits | baseline, 3 months, 6 months, 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures.
Associated costs of patients encountering emergency room (ER) visits | baseline, 3 months, 6 months, 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures.
The number of patients encountering psoriasis-related procedures | baseline, 3 months, 6 months, 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures.
Associated costs of patients encountering psoriasis-related procedures | baseline, 3 months, 6 months, 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures.
The number of psoriasis-related physician encounters in a subgroup of patients treated with brodalumab and a matched cohort at 12 months post brodalumab initiation. | 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures
The associated costs of psoriasis-related physician encounters in a subgroup of patients treated with brodalumab and a matched cohort at 12 months post brodalumab initiation. | 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures
The number of hospital encounters in a subgroup of patients treated with brodalumab and a matched cohort at 12 months post brodalumab initiation. | 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures
The associated costs of hospital encounters in a subgroup of patients treated with brodalumab and a matched cohort at 12 months post brodalumab initiation. | 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures
The number of emergency room (ER) visit encounters in a subgroup of patients treated with brodalumab and a matched cohort at 12 months post brodalumab initiation | 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures
The associated costs of emergency room (ER) visit encounters in a subgroup of patients treated with brodalumab and a matched cohort at 12 months post brodalumab initiation | 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures
The number of psoriasis-related procedures encounters in a subgroup of patients treated with brodalumab and a matched cohort at 12 months post brodalumab initiation. | 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures
The associated costs of psoriasis-related procedures encounters in a subgroup of patients treated with brodalumab and a matched cohort at 12 months post brodalumab initiation. | 12 months
  Healthcare encounters include: psoriasis-related physician, hospital and emergency room (ER) visits, as well as psoriasis-related procedures

CONTACTS AND LOCATIONS:
Overall Officials: Martin Barbeau, Study Director — Bausch Health
Locations (42):
- Canada (42):
  - CARE Site 42, Calgary, Alberta
  - CARE Site 26, Calgary, Alberta
  - CARE Site 15, Calgary, Alberta
  - CARE Site 18, Edmonton, Alberta
  - CARE Site 41, Edmonton, Alberta
  - CARE Site 21, Edmonton, Alberta
  - CARE Site 37, Edmonton, Alberta
  - CARE Site 28, Sherwood Park, Alberta
  - CARE Site 31, Vancouver, British Columbia
  - CARE Site 36, Winnipeg, Manitoba
  - CARE Site 12, Winnipeg, Manitoba
  - CARE Site 35, Saint Johns, Newfoundland and Labrador
  - CARE Site 11, Ajax, Ontario
  - CARE Site 05, Barrie, Ontario
  - CARE Site 06, Greater Sudbury, Ontario
  - CARE Site 20, Guelph, Ontario
  - CARE Site 14, Hamilton, Ontario
  - CARE Site 24, Hamilton, Ontario
  - CARE Site 23, London, Ontario
  - CARE Site 22, London, Ontario
  - CARE Site 09, London, Ontario
  - CARE Site 33, Markham, Ontario
  - CARE Site 44, Mississauga, Ontario
  - CARE Site 51, Niagara Falls, Ontario
  - CARE Site 48, North York, Ontario
  - CARE Site 27, Oshawa, Ontario
  - CARE Site 13, Richmond Hill, Ontario
  - CARE Site 49, Toronto, Ontario
  - CARE Site 16, Toronto, Ontario
  - CARE Site 32, Whitby, Ontario
  - CARE Site 38, Drummondville, Quebec
  - CARE Site 07, Laval, Quebec
  - CARE Site 50, Laval, Quebec
  - CARE Site 04, Montreal, Quebec
  - CARE Site 46, Québec, Quebec
  - CARE Site 30, Québec, Quebec
  - CARE Site 17, Québec, Quebec
  - CARE Site 52, Saint-Charles-Borromée, Quebec
  - CARE Site 39, Saint-Jérôme, Quebec
  - CARE Site 47, Sherbrooke, Quebec
  - CARE Site 40, Westmount, Quebec
  - CARE Site 03, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided